CLINICAL TRIAL: NCT01244737
Title: Phase 2 Study of [18F]FLT for PET Imaging of Brain Tumors in Children
Brief Title: FLT-PET Imaging of Brain Tumors in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Frederick Daniel Grant (Other)
Collaborators: Dana-Farber Cancer Institute (Other)
Responsible Party: Sponsor-Investigator, Frederick Daniel Grant, Assistant Professor in Radiology, Boston Children's Hospital
Organization: Boston Children's Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: IND 104365; R01FD003718 (FDA)
Record Dates: First submitted 2010-10-29; First posted 2010-11-19 (Estimated); Results first posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-06

CONDITIONS: Brain Neoplasms
Keywords: Brain neoplasms; Children; Positron-Emission Tomography; 18F-FLT
MeSH Terms: conditions — Brain Neoplasms | interventions — alovudine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- New diagnosis of brain tumor (Experimental): In children with a new diagnosis of central nervous system tumor, a PET scan will be performed using [18F] FLT.
  Interventions: Drug: [18F] FLT
- Possible recurrent brain tumor (Experimental): In children in whom there is concern for recurrent central nervous system tumor, a PET scan will be performed using [18F] PET.
  Interventions: Drug: [18F] FLT
- Brain tumor response to chemotherapy (Experimental): In children with a newly diagnosed central nervous system tumor who will be treated with post-operative chemotherapy, a PET scan will be performed using [18F] FLT before the start and after two cycles of chemotherapy.
  Despite much effort and working with referring physicians at multiple hospitals, enrollment in this arm remained low, and it seemed unlikely that meaningful enrollment would be accomplished. A revised study plan was submitted to the granting agency and FDA, and this arm was closed to further enrollment.
  Interventions: Drug: [18F] FLT

INTERVENTIONS:
Drug: [18F] FLT — [18F] FLT, intravenous, at a dose of 0.15 mCi/kg once before a PET scan
  Other Names: 3'-deoxy-3'-[F-18] fluorothymidine; [18F] fluorothymidine

SUMMARY:
Brain tumors are the leading cause of death from solid tumors in children. Tumor imaging is important in the management of these tumors, but current imaging methods have limitations in providing the necessary information for optimal treatment of these patients. The goal of this study is to evaluate the potential utility of positron emission tomography (PET) with 3'-deoxy-3'-[F-18] fluorothymidine (18F-FLT) in the medical management of brain tumors in children. Funding source - FDA Office of Orphan Product Development (OOPD)

DETAILED DESCRIPTION:
Although pediatric central nervous system tumors are rare, they are a significant contributor to morbidity and mortality in children. Tumor staging, detecting recurrent tumor, and assessing the response to therapy are critical in the treatment of brain tumors, but current imaging methods have major limitations in providing such information. The objective of this study is to validate 3'-deoxy-3'-[F-18] fluorothymidine (18F-FLT) as a measure of tumor proliferation and to demonstrate the utility of 18F-FLT as a PET imaging agent in children with central nervous system tumors. The proposed studies will evaluate 18F-FLT PET in three groups:

1. Children with a new diagnosis of central nervous system tumor.
2. Children in whom conventional imaging has raised concern for possible recurrence of a central nervous system tumor.
3. Children receiving post-operative chemotherapy for a central nervous system tumor.

In these three groups, correlation of 18F-FLT uptake with tumor histopathology and patient outcome will be used to assess the utility of 18F-FLT for grading tumors at diagnosis, for accurate identification of tumor recurrence, and for early assessment of the response to chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* age 21 years or less
* capable of achieving imaging without need for sedation or anesthesia (typically age 8 years or greater, but there is no lower limit for age for eligibility)
* Karnofsky Performance Status of 50 or greater in subjects age 12 years or greater, for age less than 12 years a Lansky play scale of 50% or greater
* Patients receiving steroids and/or anti-seizure medications are eligible

Exclusion Criteria:

* clinically active infection
* pregnancy or breast-feeding
* serious intercurrent medical illness
* require emergency surgical intervention that would be inappropriately delayed by FLT-PET imaging

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2023-02-05 (Actual); Study Completion 2023-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick D Grant, MD, Principal Investigator — Children's Hospital, Boston, Harvard Medical School
Locations (1):
- Children's Hospital, Boston, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
No current plans to share individual participant data

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential participants were identified by clinicians participating in their care.
Pre-assignment Details: Participants were assigned to one of three arms, depending on clinical presentation: 1) Clinical concern for new brain tumor, 2) Clinical concern for recurrent brain tumor, or 3) Planned initiation of new chemotherapy for a known brain tumor
Groups:
- Brain Tumor Response to Chemotherapy: In children with a newly diagnosed central nervous system tumor who will be treated with post-operative chemotherapy, a PET scan will be performed using [18F] FLT before the start and after two cycles of chemotherapy.
  Despite much effort and working with referring physicians at multiple hospitals, enrollment in this arm remained low, and it seemed unlikely that meaningful enrollment would be accomplished. A revised study plan was submitted to the granting agency and FDA, and this arm was closed to further enrollment.
  [18F] FLT: [18F] FLT, intravenous, at a dose of 0.15 mCi/kg once before a PET scan
Period: Overall Study
Arm/Group | New Diagnosis of Brain Tumor | Possible Recurrent Brain Tumor | Brain Tumor Response to Chemotherapy
Started | 16 | 28 | 6
Successful Completion of FLT-PET | 14 | 26 | 5
Surgery Within 30 Days of FLT-PET | 13 | 8 | 0
Surgical Pathology Demonstrated Evaluable Brain Tumor | 11 | 7 | 0
MIB Immunohistology Available | 8 | 5 | 0
Completed | 8 | 5 | 0
Not Completed | 8 | 23 | 6
Not completed — Physician Decision | 2 | 18 | 5
Not completed — Radiopharmaceutical FLT (18F-fluorothymidine) unavailable to perform PET scan before surgery | 1 | 1 | 0
Not completed — Surgical pathology did not confirm evaluable brain tumor | 2 | 1 | 0
Not completed — MIB immunopathology results not available | 3 | 2 | 0
Not completed — PET data failure | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- New Diagnosis of Brain Tumor: In children with a new diagnosis of central nervous system tumor, a PET scan will be performed using [18F] FLT.
  [18F] FLT: [18F] FLT, intravenous, at a dose of 0.15 milliCurie (mCi)/kg once before a PET scan
- Total: Total of all reporting groups
Arm/Group | New Diagnosis of Brain Tumor | Possible Recurrent Brain Tumor | Brain Tumor Response to Chemotherapy | Total
Number analyzed (Participants) | 16 | 28 | 6 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16 | 27 | 6 | 49
  Between 18 and 65 years | 0 | 1 | 0 | 1
  >=65 years | 0 | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 1 | 15 | 1 | 17
  Male | 13 | 11 | 4 | 28
  Other/ Not recorded | 2 | 2 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 6 | 1 | 9
  Not Hispanic or Latino | 12 | 19 | 4 | 35
  Unknown or Not Reported | 2 | 3 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 3 | 3 | 2 | 8
  White | 9 | 16 | 3 | 28
  More than one race | 2 | 3 | 0 | 5
  Unknown or Not Reported | 2 | 2 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 16 | 28 | 6 | 50
Brain Tumor classification [Count of Participants; unit: Participants] — derived from major categories from: World Health Organization (WHO) Classification of Brain Tumors, 5th edition (2021)
  Participants
    Gliomas, Glioneuronal, and Neuronal Tumors | 11 | 18 | 5 | 34
    Embryonal Tumors (including former PNET) | 1 | 7 | 1 | 9
    Pineal Tumors | 1 | 0 | 0 | 1
    Germ Cell Tumors (Teratoma) | 0 | 1 | 0 | 1
    Hematolymphoid Tumors (Lymphoma) | 1 | 0 | 0 | 1
    Non-neoplastic Process/No Diagnosis | 2 | 2 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: [18F] Fluorothymidine ([18F]-FLT) Uptake as a Marker of Cellular Proliferation
Description: [18F] FLT uptake, as determined by pre-operative positron emission tomography (PET) imaging, will be compared to histological markers of cellular proliferation in the resected brain tumor. This will be performed in three groups of subjects (3 arms): (1)children with newly diagnosed central nervous system tumors, (2) children in whom there is concern for recurrence of central nervous system tumor,(3) children with central nervous system tumors that are treated with post-operative chemotherapy.
Time Frame: on average 1 week
Population: Participants were evaluable if brain tumor surgery was performed within 30 days of the FLT-PET scan, if surgical pathology confirmed the diagnosis of brain tumor, and the results of tissue immunohistology were available. On the brain PET scan, tumor uptake of FLT was assessed by SUVmax, the standard clinical measure of tracer uptake, and tumor proliferation was assessed as the fraction of cells with positive MIB immunostaining
Measure: Mean (Full Range); unit: SUV max
Arm/Group | New Diagnosis of Brain Tumor | Possible Recurrent Brain Tumor
Number analyzed (Participants) | 8 | 5
SUV max | 1.57 [0.12 to 4.00] | 3.00 [1.54 to 4.00]
Statistical Analysis 1: Comparison: New Diagnosis of Brain Tumor vs Possible Recurrent Brain Tumor; This is a diagnostic test of FLT uptake (SUV max) as a predictor of cellular proliferation (MIB) and is performed as an analysis of correlation using each evaluable participant enrolled in either Arm 1 (New Diagnosis) or Arm 2 (Possible recurrent tumor). The groups (Arm 1 and Arm 2) provide pathways for enrollment. Correlation between the two measures of outcome (SUV max and MIB) is evaluated; Test type: Other; p < 0.001, Regression, Linear — The a priori threshold for statistical significance was < 0.05; Pearson correlation co-efficient = 0.80

2. Primary Outcome: MIB Positive (Percent)
Description: On pathological specimens, tumor proliferation was assessed as the fraction of cells with positive MIB immunostaining
Time Frame: 30 days
Population: Participants in Arm 3 (Brain tumor response to chemotherapy) were not expected to undergo surgery during their chemotherapy. Therefore, they did have FLT-PET, but no assessment for tumor proliferation (percent MIB positive) was performed.
Measure: Mean (Full Range); unit: percent positive cells
Groups:
- New Diagnosis of Brain Tumor: In children with a new diagnosis of central nervous system tumor and who undergo surgery within 30 days of FLT-PET, surgical pathological specimens will be analyzed using immunohistologic staining with MIB as a measure of tumor proliferation
- Possible Recurrent Brain Tumor: In children in whom there is concern for recurrent central nervous system tumor and who undergo surgery within 30 days of FLT-PET, surgical pathological specimens will be analyzed using immunohistologic staining with MIB as a measure of tumor proliferation
Arm/Group | New Diagnosis of Brain Tumor | Possible Recurrent Brain Tumor
Number analyzed (Participants) | 8 | 5
percent positive cells | 17.3 [0.9 to 59.4] | 32.8 [4.3 to 89]

3. Secondary Outcome: Biodistribution of [18F]FLT
Description: The distribution, localization, and kinetics of localization of [18F] FLT will be assessed by FLT-PET in 12 subjects.
Time Frame: 6 hours
Population: Saved PET scan data has not been retrievable or usable due to 1) storage/format incompatibility among PET cameras from different vendors, 2) lack of interoperablity among different generations of cameras from the same vendor, and 3) backup data in institutional radiology archiving systems is not universally available for retrieval for quantitative image analysis. To date, working with camera vendors and software developers has been unsuccessful in overcoming this problem.
Arm/Group | New Diagnosis of Brain Tumor | Possible Recurrent Brain Tumor | Brain Tumor Response to Chemotherapy
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Preliminary Evaluation of Clinical Utility of [18F] FLT PET
Description: In individuals with a diagnosed primary brain tumor in whom therapy will include chemotherapy,.[18F] FLT uptake, as determined by positron emission tomography (PET) imaging, will assessed before and after two cycles of chemotherapy. Response will be determined by comparing the FL uptake before and after therapy.
Time Frame: 3 months
Population: Despite much effort and working with referring physicians at multiple hospitals, enrollment in this arm remained low and participant completion of the entire protocol was low. As it seemed unlikely that meaningful enrollment would be accomplished, a revised study plan was submitted to the granting agency and FDA, and this arm was closed to further enrollment. Due to the small number of participants completing the protocol, FLT uptake was assessed, but clinical outcome was not evaluated.
Measure: Mean (Full Range); unit: SUV max
Arm/Group | Brain Tumor Response to Chemotherapy
Number analyzed (Participants) | 6
SUV max
  FLT uptake pre-therapy: number analyzed (Participants) | 5
  FLT uptake pre-therapy | 0.85 [0 to 1.53]
  FLT uptake post-therapy: number analyzed (Participants) | 3
  FLT uptake post-therapy | 0.47 [0 to 1.13]
Statistical Analysis 1: Comparison: Brain Tumor Response to Chemotherapy; Test type: Other — Paired T-test to assess change in FLT uptake (SUV max) with chemotherapy; p = 0.04, t-test, 2 sided — The a priori threshold for statistical significance was < 0.05

ADVERSE EVENTS:
Time Frame: 1 week
Description: Systemic: Complete blood count and renal/liver labs before and after each FLT-PET. One week after FLT-PET, medical record review for adverse events.
  Non-systemic: Referring clinicians inform study team of severe adverse events. Review: Adverse events reported to the Institutional Review Board (IRB) using current institutional procedures. Two severe adverse events reviewed by the IRB were judged to be consistent with the underlying brain tumor and associated therapy, and not due to FLT-PET.
Arm/Group | New Diagnosis of Brain Tumor | Possible Recurrent Brain Tumor | Brain Tumor Response to Chemotherapy
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/28 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/16 | 2/28 | 0/6
Other Adverse Events (participants affected / at risk) | 1/16 | 3/28 | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | New Diagnosis of Brain Tumor (N=16) | Possible Recurrent Brain Tumor (N=28) | Brain Tumor Response to Chemotherapy (N=6)
intracranial tumor hemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — intracranial tumor hemorrhage
reversible posterior leukoencephalopathy sydrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | New Diagnosis of Brain Tumor (N=16) | Possible Recurrent Brain Tumor (N=28) | Brain Tumor Response to Chemotherapy (N=6)
urticarial rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — urticaria
anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Arm 3: Despite much recruitment effort, enrollment in this arm remained low, and it seemed unlikely that meaningful enrollment would be accomplished. A revised study plan was submitted to the granting agency and FDA, and this arm was closed to further enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/37/NCT01244737/Prot_SAP_000.pdf